CLINICAL TRIAL: NCT03711084
Title: The Impact of Dietary Sweetness on Neurocognitive Responses to Visual Food Cues, Appetite and Physiological Parameters on Normal Weight Adults: a Pilot Study
Brief Title: Effects of Sweetness on Neurocognitive Responses, Glycemia and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Cargill (Industry)
Responsible Party: Principal Investigator, Nikoleta Stamataki, PhD student, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2310
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: non-nutritive sweeteners; sucrose; food-cue responses; appetite; blood glucose; energy intake
MeSH Terms: conditions — Obesity | interventions — Glucose; Sucrose; maltodextrin; Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Water (Placebo Comparator): Beverage containing either water, glucose, sucrose, maltodextrin or a natural high potency sweetener from leaf extract
  Interventions: Dietary Supplement: Water
- Natural high potency sweetener from leaf extract (Experimental): Beverage containing either water, glucose, sucrose, maltodextrin or a natural high potency sweetener from leaf extract
  Interventions: Dietary Supplement: Natural high potency sweetener from leaf extract
- Glucose (Experimental): Beverage containing either water, glucose, sucrose, maltodextrin or a natural high potency sweetener from leaf extract
  Interventions: Dietary Supplement: Glucose
- Sucrose (Experimental): Beverage containing either water, glucose, sucrose, maltodextrin or a natural high potency sweetener from leaf extract
  Interventions: Dietary Supplement: Sucrose
- Maltodextrin (Experimental): Beverage containing either water, glucose, sucrose, maltodextrin or a natural high potency sweetener from leaf extract
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Natural high potency sweetener from leaf extract — Upon arrival, participant's blood will be collected at 0 (before the consumption of the test beverage), 15, 30 and 60 min after the consumption of the drink. Participants will rate their feelings of hunger, fullness etc using VAS at 0, 15, 30 and 60 min.
  Fifteen min after the consumption of the drink, participants will complete a set of computer-based tasks designed to capture behaviour in response to food cue presentation. Thirty min after the consumption of the drink, a lunch buffet will be served and participants will be free to eat as much or as little as they like until feeling comfortably full.
  Arms: Natural high potency sweetener from leaf extract
Dietary Supplement: Glucose — Upon arrival, participant's blood will be collected at 0 (before the consumption of the test beverage), 15, 30 and 60 min after the consumption of the drink. Participants will rate their feelings of hunger, fullness etc using VAS at 0, 15, 30 and 60 min.
  Fifteen min after the consumption of the drink, participants will complete a set of computer-based tasks designed to capture behaviour in response to food cue presentation. Thirty min after the consumption of the drink, a lunch buffet will be served and participants will be free to eat as much or as little as they like until feeling comfortably full.
  Arms: Glucose
Dietary Supplement: Sucrose — Upon arrival, participant's blood will be collected at 0 (before the consumption of the test beverage), 15, 30 and 60 min after the consumption of the drink. Participants will rate their feelings of hunger, fullness etc using VAS at 0, 15, 30 and 60 min.
  Fifteen min after the consumption of the drink, participants will complete a set of computer-based tasks designed to capture behaviour in response to food cue presentation. Thirty min after the consumption of the drink, a lunch buffet will be served and participants will be free to eat as much or as little as they like until feeling comfortably full.
  Arms: Sucrose
Dietary Supplement: Maltodextrin — Upon arrival, participant's blood will be collected at 0 (before the consumption of the test beverage), 15, 30 and 60 min after the consumption of the drink. Participants will rate their feelings of hunger, fullness etc using VAS at 0, 15, 30 and 60 min.
  Fifteen min after the consumption of the drink, participants will complete a set of computer-based tasks designed to capture behaviour in response to food cue presentation. Thirty min after the consumption of the drink, a lunch buffet will be served and participants will be free to eat as much or as little as they like until feeling comfortably full.
  Arms: Maltodextrin
Dietary Supplement: Water — Upon arrival, participant's blood will be collected at 0 (before the consumption of the test beverage), 15, 30 and 60 min after the consumption of the drink. Participants will rate their feelings of hunger, fullness etc using VAS at 0, 15, 30 and 60 min.
  Fifteen min after the consumption of the drink, participants will complete a set of computer-based tasks designed to capture behaviour in response to food cue presentation. Thirty min after the consumption of the drink, a lunch buffet will be served and participants will be free to eat as much or as little as they like until feeling comfortably full.
  Arms: Water

SUMMARY:
This study aims to examine potential differences in neurocognitive responses to food-related cues, physiological and appetite responses as well as subsequent energy intake following the consumption of preloads differing in sweetness and/ or postprandial metabolic effects in healthy normal weight subjects.

DETAILED DESCRIPTION:
Excess consumption of caloric sweeteners, together with the high availability of palatable food cues are some of the factors for the alarming high rates of overweight and obesity. Although non-nutritive sweeteners (NNS) are used to decrease energy content of foods and beverages, there is an on-going debate on the relationship between NNS intake, obesity and cardiometabolic risk. Caloric sugars have a differing effect on physiological responses compared to NNS. However it is almost wholly unknown how NNS consumption affects eating behaviour and cognitive processes.

This study compares the performance on food related neurocognitive tasks following the consumption of the test preloads on 5 visits. In particular, sucrose, glucose, maltodextrin, water or a natural high potency sweetener from leaf extract will be ingested as single test agents in randomized order. Water will be used as a control for gastric distension and non-sweet, whereas maltodextrin will be used as a non-sweet control for carbohydrate content.

Participants will be asked to attend a screening visit at the Neuroscience and Psychiatry Unit of the University of Manchester on a morning after overnight fast. Participants' weight and height, fasting blood glucose and blood pressure will be measured. This will be followed by some questionnaires regarding general health status, weight and dieting history and eating behaviour.

Participants who satisfy the inclusion criteria, will be then invited to take part in the full study. This will require 5 separate visits at the University of Manchester, which will be scheduled between 11.30 and 13.30. Participants will have to attend these visits after having fasted for 3-4 hours and will be asked to have their regular breakfast in the morning before the testing session, and then not eat or drink anything else for 3-4 hours until they come in the lab for the testing session. Water will be allowed up to 1 hour prior to your testing session. Prior to each testing session participants will be asked to have the same breakfast, and they will have to provide a picture of the breakfast each time to ensure compliance.

The 5 visits correspond to 5 test beverages, both the participants and the investigators are blinded to the study treatments. Blood will be collected at 0 (before the consumption of the test beverage), 15, 30 and 60 min after the consumption of the drink. Participants will also be asked to rate their feeling of hunger, fullness etc using visual analogue scales (VAS) at the same time points 0, 15, 30 and 60 min.

Fifteen min after the consumption of the drink, participants will complete a set of computer-based tasks. They are designed to capture behaviour in response to food cue presentation. This will last approximately 15 min.

Thirty min after the consumption of the drink, a lunch buffet will be served and participants will be free to eat as much or as little as they like until feeling comfortably full. Each session is anticipated to last for approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years
* BMI between 18.5-24.9 kg/m2
* DEBQ for restraint eating ≤ 3
* Healthy - general good health
* Currently not taking any medication (other than females taking the oral contraceptives)
* Normal or corrected vision
* Regular breakfast eaters (≥5 times per week)
* Stable weight, ≤ 5 kg last 12 months
* Fasting blood glucose ≤6.0 mmol/L
* No self-reported food allergy or intolerance to foods supplied during the study
* The participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The participant is able to read, comprehend and record information written in English.
* A signed and dated written informed consent is obtained from the participant.

Exclusion Criteria:

* Age under 18 years or over 40 years old.
* BMI ≥25 kg/m2 and <18.5kg/m2
* Subjects who are currently on a diet
* Subjects who follow special diets for weight maintenance, such as Atkins Diet, Weight Watchers, gluten-free diet, The Zone diet, Vegetarian Diet, Raw Food Diet etc.
* Subjects having breakfast fewer than 5 times per week.
* Vegetarians, vegans.
* Presence of any chronic condition requiring medication that might affect our results (e.g. diabetes, mental diseases, gastrointestinal diseases)
* Subjects with eating disorders (binge eating disorder, bulimia etc)
* Subjects who are currently experiencing anxiety or depression.
* Subjects who do not have normal vision and do not correct it with glasses or contact lenses.
* Participants who drink more than the NHS guidelines (14 units per week)
* Female participants who are, or may be, pregnant, or currently lactating.
* Subjects who regularly consume dietary supplements for weight loss, muscle building etc.
* Subjects who have aversions to foods related with the study.
* Subjects with food allergies or intolerance related with the foods/ drinks of the study.
* Habitual NNS consumers, >1 can of diet beverage or >1 table packet of sweeteners per week.
* Fasting blood glucose measured > 6 mmol/L at screening visit, according to diabetes.co.uk recommendations.
* The participant cannot read, comprehend and record information written in English.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Energy intake | 1 hour
  Examine how the consumption of sweet vs. non- sweet and energy-containing vs. non-energy containing preloads affects energy intake (kcal) in healthy lean individuals.
Appetite ratings | 1 hour
  Examine how the consumption of sweet vs. non- sweet and energy-containing vs. non-energy containing preloads affects appetite ratings (VAS scales) in healthy lean individuals.
Food-cue responses | 1 hour
  Examine how the consumption of sweet vs. non- sweet and energy-containing vs. non-energy containing preloads affects food-cue responses (reaction times) in healthy lean individuals.
Blood glucose levels | 1 hour
  Examine how the consumption of sweet vs. non- sweet and energy-containing vs. non-energy containing preloads affects blood glucose levels (mmol/L) in healthy lean individuals.

SECONDARY OUTCOMES:
Hedonic ratings | 1 hour
  Examine how participants rate the hedonic attributes of the test beverages (Sweetness, pleasantness, etc) and the meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stamataki NS, Scott C, Elliott R, McKie S, Bosscher D, McLaughlin JT. Stevia Beverage Consumption prior to Lunch Reduces Appetite and Total Energy Intake without Affecting Glycemia or Attentional Bias to Food Cues: A Double-Blind Randomized Controlled Trial in Healthy Adults. J Nutr. 2020 May 1;150(5):1126-1134. doi: 10.1093/jn/nxaa038. PMID 32125421